CLINICAL TRIAL: NCT04795271
Title: Biomechanical Study of Patients With Diabetic Foot for the Establishment of a Preventive Orthopedic Treatment Protocol for Major Complications
Brief Title: Biomechanical Study and Orthopedic Treatment Prevent in People With Diabetic Foot
Acronym: FOOTprevent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Valencia (Other)
Collaborators: Instituto de Investigacion Sanitaria INCLIVA (Other)
Responsible Party: Principal Investigator, Constanza San Martín, Researcher, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020/028
Record Dates: First submitted 2021-03-09; First posted 2021-03-12 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Diabetic Foot
Keywords: Diabetic foot; Biomechanical assessment; Orthopedic treatment
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: All participants will receive personalized orthopedic treatment, depending on the plantar discharge needs that each patient needs. This treatment may include the use of an insole or insole and orthopedic footwear.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orthopedic treatment (Experimental): Participants who are referred for orthopedic treatment as indicated by the treating traumatologist or rehabilitating doctor will be evaluated and treated by one of the three orthopedists participating in this study.
  After the orthopedic evaluation, the professional will determine the most suitable insole according to the plantar discharge needs required by the patient. The intervention in the insole can include modifications or corrections at the forefoot, midfoot, or hindfoot. The material used in each insole will also be specified. When the insole requires many modifications and raises the height of the subject's foot, the use of orthopedic footwear will also be added to prevent pressure on the dorsum of the foot that could be caused by normal footwear.
  Interventions: Other: Orthopedic intervention

INTERVENTIONS:
Other: Orthopedic intervention — In each custom insole, modifications can be included in the following aspects according to the requirements of each participant :
  1. Forefoot specifications: a) Retrocapital bar, b) Retrocapital support, c) Claw toe correction element, d) Pronating wedge, e) Supinator wedge, f) Metatarsal head pad, g) Selective perforations in the insole, h) Others.
  2. Midfoot specifications: a) Internal arch, b) External arch, c) Full support, d) Excavations, e) Others.
  3. Hindfoot specifications: a) Heel cup, b) Supinator wedge, c) Pronating wedge, d) Lifter, e) Cup, f) Others.
  4. Insole type and lining material
  5. Materials of the added corrections
  6. Insole base: a) soft ethylene vinyl acetate (eva), b) semi-soft eva, c) hard eva, d) rubber, e) cuerolite.

SUMMARY:
Spain is the country with the second-highest rate of population amputation due to the development of ulcers, behind the United States, where 2 out of 3 non-traumatic amputations derive from diabetes. This is why the main objective of this project is to establish a study protocol for alterations in plantar pressures and gait abnormalities in diabetic patients, parallel to the preventive orthopedic treatment of major complications such as Charcot's foot, ulcers in the plantar support surface, and amputations. The study methodology will be based on the evaluation prior to the personalized orthopedic treatment for each patient and the evaluation after the orthopedic treatment, specifically at one week, one month, three months, and six months after the treatment. At each evaluation time, plantar pressure and reaction forces during walking and local infrared thermography will be analyzed. In the basal and final evaluation at six months, the muscular strength and range of motion of the lower limbs will also be evaluated. The orthopedic intervention is personalized to the requirements of the patients and is based on the use of an insole with the possible inclusion of orthopedic footwear in order to reduce plantar pressure.

DETAILED DESCRIPTION:
Background

Diabetic foot is the syndrome characterized by tissue changes (skin, joint, and/or bone) of the feet of diabetic patients as a result of peripheral neuropathy induced by high glucose levels, which can be aggravated by the coexistence of microcirculation alterations blood and whose production involves micro-traumas as a result of support during walking. When tissue repair or regeneration mechanisms are not effective, these initial lesions can evolve into ulcerations, superficial and/or deep infections, osteomyelitis or dislocations of the foot joints (Charcot's foot), with serious consequences for the patient such as limb amputation, whose costs for Public Health are high. It should be taken into account that Spain is the country with the second-highest rate of population amputation due to the development of ulcers, behind the United States, where 2 out of 3 non-traumatic amputations derive from diabetes.

This is why the main objective of this project is to establish a study protocol for alterations in plantar pressures and gait abnormalities in diabetic patients, parallel to the preventive orthopedic treatment of major complications such as Charcot's foot, ulcers in the plantar support surface, and amputations.

As specific objectives proposed are the following:

1. To evaluate and objectify the clinical and biomechanical alterations of people with Diabetic foot before orthopedic treatment.
2. To analyze the effects of immediate orthopedic treatment in the medium and long term in people with Diabetic foot through biomechanical and clinical parameters.
3. To determine if the biomechanical analysis influences the decisions of the trauma doctors and rehabilitators treating the study participants.

Methodology

1. General organization

   The traumatologists (3) and the rehabilitation physician (1) who are part of the research team of the study will recruit the participants from the medical consultation that they maintain at the participating hospital in this study. Through compliance with the inclusion criteria, patients will be invited to enter the study. Those who agree to participate will sign the corresponding informed consent and will be referred for the baseline evaluation. The assessment times are as follow:
   * Baseline evaluation after signing the informed consent Orthopedic evaluation and implementation of orthopedic treatment
   * Evaluation at one week after starting orthopedic treatment
   * Evaluation at one month after starting orthopedic treatment
   * Evaluation at three months after starting orthopedic treatment
   * Evaluation at six months after starting orthopedic treatment
2. Session assessment

In each of the evaluation sessions mentioned above, the following data and outcomes will be recorded:

2.1 Clinical assessment: The clinical evaluation will consist of determining the main anatomical variables that describe the foot of the participants. These variables will be determined in consultation with a traumatologist or rehabilitation physician at the time of patient recruitment. It will be determined: a) arch of the foot: this polytomous variable determines whether the patient has cavus or flat feet; b) Moreau-Costa-Bartani angle (º); c) Astragalus-calcaneus angle (º); d) Hindfoot alignment: this polytomous variable indicates whether the patient has a valgus, varus or neutral hindfoot; e) Toe position: this polytomous variable describes whether the subjects present any of the toes in hyperextension of the metatarsophalangeal joint with proximal interphalangeal and distal interphalangeal flexion (claw), or have normal anatomy and position; f) Posterior tibial pulse: explores the posterior tibial artery, palpated at the ankle at the level of the posterior area of the external malleolus (internal retro-malleolar canal); g) Pedic pulse: explores the pediatric artery, palpates at the level of the dorsal aspect of the foot between the extensor tendons of the 1st and 2nd toes, it can also frequently be palpated between the 2nd and 3rd.

2.2 Anthropometric assessment: A series of essential preliminary measurements will be carried out for the normalization of biomechanical data and its subsequent comparison between subjects. The following will be evaluated: a) Weight measurement on the force platform (Kg); b) Height measurement on stadiometer (Cm); c) Measurement of the arm, leg, and waist contour measured with a tape measure (Cm); d) Measurement of BMI, body water percentage (%) and body fat percentage (%) will be extracted with an analytical scale.

2.3 Range of motion assessment: Joint range measurements will be measured with the NeDSGE 4.1 electronic goniometer and NedDiscapacidad / IBV V4.1.1 software (Institute of Biomechanics of Valencia, Spain) that allows data to be recorded and stored digitally. a) Measurements in the hip joint: flexion and extension, internal and external rotation, abduction and adduction; b) Measurements in the knee joint: flexion and extension; c) Measurements in the ankle joint: dorsal flexion, plantar flexion, inversion, and eversion.

2.4 Muscular strength assessment: To evaluate the degree of muscular force (Newton), an electronic dynamometer NedDFM/IBV and software NedDiscapacidad/IBV V4.1.1 will be used (Institute of Biomechanics of Valencia, Spain), which allows the evaluation and recording of muscular force performed digitally. Three measurements of maximum strength will be obtained for each gesture, without these differing by more than 10% from each other. a) Muscle strength measured from the hip flexors, extensors, abductors, adductors, and internal and external rotators; b) Measured muscle strength of the knee flexor and extensor muscles; c) Muscle strength measured from the plantar flexor and dorsiflexor muscles of the foot.

2.5 Assessment of speed and ground reaction forces during walking: During the evaluation, the patient should walk in a 10-meter long corridor, in a straight line at a comfortable or self-selected speed. Two dynamometric platforms will be used to record the ground reaction forces during the tread, and two pairs of infrared sensors to record the speed. The software we use for this evaluation is AMH / IBV 4.0.4. The outcomes obtained from the gait analysis are; a) Walking speed (m / s); b) Support time (s): proportion of total time spent during the support phase. Initiated in the contact of a hindfoot and ending in the detachment of the toes of the same foot. c) Braking force: minimum registered anterior-posterior ground reaction force corresponding to heel strike (N), d) Propulsive force: maximum registered anterior-posterior ground reaction force corresponding to takeoff (N), e) Swing force: minimum registered vertical ground reaction force occurring during contralateral foot oscillation (N), f) Push-off force: second highest register of the vertical component of ground reaction force that occurs between heel-off and toe-off (N).

2.6 Assessment of plantar pressure during standing position and walking: The evaluation of plantar pressures will be carried out during standing position and walking in a straight line at a comfortable speed. The measuring instrument consists of instrumented insoles with pressure sensors, which will go inside the patient's footwear. The software used is the Biofoot/IBV Version 6b. The corridor to be covered by the patient is 10 meters, on which they can be recorded in five and six strides according to the different lengths of the participants' stride. The main outcomes obtained from plantar pressure assessment are: a) Support time (s): total duration of foot contact with the ground; b) cadence (step / min); c) Maximum pressure (%): maximum pressure value obtained in the analyzed area; d) Maximum pressure time (%): moment in the support phase in which the maximum pressure value is reached, expressed as a percentage of time in relation to the total duration of the footfall; e) Maximum mean pressure (kpa): Maximum value of the mean pressure of the analyzed area expressed in kilopascals; f) Maximum time of the average pressure (%): instance of the support phase in which the maximum of the average pressure occurs, expressed as a percentage of time in relation to the total duration of the tread; g) Integral of Mean Pressure: area under the curve described by mean pressure over time.

2.7 Thermographic assessment: Thermographic images were recorded before and after of gait measurements. Before walking, the change in temperature was also observed when a cold stimulus was applied to the plantar of both foot. All thermographic images were recorded digitally by a thermography camera with an infrared resolution of 320×240 pixels, thermal sensitivity <0.05 °C, and accuracy of ±2 °C (FLIR E60, FLIR, Wilsonville, Oregon, USA). A black body (BX-500 IR Infrared Calibrator, CEM, Shenzhen, China) was used before the study to ensure a correct calibration of the camera. The camera was positioned 1 m far from the subjects and kept perpendicular to body areas of interest. Images were recorded in a controlled environment (e.g. light and temperature controlled room) with no person (apart from the infrared operator and the participant) or equipment in a range of 5 m that could disturbed in the measure. An anti-reflective panel was used behind the participant to minimize effects from infrared radiation reflected by the participant in the wall. Images were stored for offline analysis using a commercial software (Thermacam Researcher Pro 2.10 software, FLIR, Wilsonville, Oregon, USA). All images were processed using an emissivity factor of 0.98 to obtain skin temperatures, and for all measures, air temperature, humidity, and reflected temperature were informed in the camera setup using a weather station (Digital thermo-hygrometer, TFA Dostmann, Wertheim-Reicholzheim, Germany).

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic polyneuropathy
* Metatarsalgia with hyperkeratosis and/or claw fingers with diabetic polyneuropathy
* Support abnormalities in the coronal plane (supination/pronation)
* Plantar ulcers secondary to alterations in evolving and healed plantar pressures
* Charcot foot postoperative

Exclusion Criteria:

* Peripheral arterial disease (absence of distal pulses or ischemia)
* Active osteomyelitis
* Patients with prostheses after amputation
* Patients who travel mainly in a wheelchair due to gait abnormalities associated with other diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in the maximum plantar pressure (kPa) | 6 months
  Maximum plantar pressure (kPa) detected in the baseline measurement and after 6 months of the use of orthopedic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Forriols Brocal, PhD., Principal Investigator — Orthopedic Surgery and Traumatology Service of the University Clinical Hospital of Valencia, Spain.
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
All data obtained through this study will be shared with the scientific community and with other researchers through scientific publications generated from this study. The principal investigators are totally open to answering questions and providing data that have previously been published if other investigators so request.